CLINICAL TRIAL: NCT06258265
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel Design Thorough QT Study With Nested Crossover to Investigate the Potential of TAK-279 to Prolong the QTc Interval in Adult Healthy Subjects
Brief Title: A Study of TAK-279 in Healthy Adults on the Effect on ECG Measurements
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-279-1001
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Therapeutic Dose Cohort: TAK-279 + TAK-279 Placebo + Moxifloxacin Placebo (Experimental): Participants will receive TAK-279 Dose 1 and matching placebo, capsules, once daily (QD) on Days 1 to 7 with moxifloxacin matching placebo, capsule, once on Days 1 and 8.
  Interventions: Drug: TAK-279; Drug: TAK-279 Placebo; Drug: Moxifloxacin Placebo
- Cohort 2, Supratherapeutic Dose Cohort: TAK-279 + Moxifloxacin Placebo (Experimental): Participants will receive TAK-279 Dose 2, capsules, QD on Days 1 to 7 with moxifloxacin matching placebo, capsule once on Days 1 and 8.
  Interventions: Drug: TAK-279; Drug: Moxifloxacin Placebo
- Cohort 3A, Control Cohort: Moxifloxacin + TAK-279 Placebo + Moxifloxacin Placebo (Experimental): Participants will receive moxifloxacin Dose 3, over-encapsulated tablet on Day 1 with TAK-279 matching placebo, QD on Days 1 to 7 and moxifloxacin placebo, capsule, once on Day 8.
  Interventions: Drug: TAK-279 Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Cohort 3B, Control Cohort: TAK-279 Placebo + Moxifloxacin Placebo + Moxifloxacin (Experimental): Participants will receive moxifloxacin matching placebo, capsule on Day 1 with TAK-279 matching placebo, QD on Days 1 to 7 and moxifloxacin Dose 3, over-encapsulated tablet, once on Day 8.
  Interventions: Drug: TAK-279 Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsule.
  Arms: Cohort 1, Therapeutic Dose Cohort: TAK-279 + TAK-279 Placebo + Moxifloxacin Placebo; Cohort 2, Supratherapeutic Dose Cohort: TAK-279 + Moxifloxacin Placebo
Drug: TAK-279 Placebo — TAK-279 matching placebo capsule.
  Arms: Cohort 1, Therapeutic Dose Cohort: TAK-279 + TAK-279 Placebo + Moxifloxacin Placebo; Cohort 3A, Control Cohort: Moxifloxacin + TAK-279 Placebo + Moxifloxacin Placebo; Cohort 3B, Control Cohort: TAK-279 Placebo + Moxifloxacin Placebo + Moxifloxacin
Drug: Moxifloxacin — Moxifloxacin over-encapsulated tablet.
  Arms: Cohort 3A, Control Cohort: Moxifloxacin + TAK-279 Placebo + Moxifloxacin Placebo; Cohort 3B, Control Cohort: TAK-279 Placebo + Moxifloxacin Placebo + Moxifloxacin
Drug: Moxifloxacin Placebo — Moxifloxacin matching placebo capsule.

SUMMARY:
The main aim of this study is to find out how more than one dose of TAK-279 changes the heart-rate corrected QT (QTc) interval of healthy adults. A QTc interval is a measurement on an electrocardiogram (ECG) and shows the time when the heart contracts until it finishes relaxing. Other aims are to learn about the effect of several doses of TAK-279 on other ECG measurements of healthy adults, how the body of a healthy adult processes TAK-279 and moxifloxacin (pharmacokinetics), and to learn about the side effects of TAK-279 and how well it is tolerated when given to healthy adults.

The participants will be given TAK-279 and moxifloxacin or a placebo for 7 days.

During the study, participants will need to stay at the clinic for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.
2. Healthy, adult, male or female, 18-55 years of age, inclusive, at the screening visit.
3. Female participants of childbearing potential and non-sterilized male participants must follow protocol specified contraception guidance as described in protocol.
4. Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first baseline cardiodynamic measurement (Day -1) based on participant self-reporting.
5. BMI greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilograms per meter square (kg/m^2) at the screening visit.
6. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and electrocardiograms (ECGs), as deemed by the Investigator or designee, including the following:

   * Supine blood pressure is >=90/40 millimeter of mercury (mmHg) and <=140/90 mmHg at the screening visit.
   * Supine pulse rate is >=40 beats per minute (bpm) and <=99 bpm at the screening visit.
   * QTc using Fridericia's formula (QTcF) interval is <=450 milliseconds (msec) (males) and <=460 msec (female) at the screening visit.
   * QRS interval <=110 msec at the screening visit (if >110 msec, result will be confirmed by a manual over read).
   * PR interval <=220 msec at the screening visit.
   * eGFR >=80 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) at the screening visit.
   * Liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin <=upper limit of normal (ULN) at the screening visit and at check-in.
   * Creatine phosphokinase (CPK) <=ULN at the screening visit and at check-in.
   * Amylase and lipase <=ULN at the screening visit and at check-in.
   * No clinically significant hypokalemia, hypomagnesemia, or other electrolyte abnormalities at the screening visit.
7. Able to swallow multiple capsules.

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to first baseline cardiodynamic measurement (Day -1), as assessed by the Investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to first baseline cardiodynamic measurement (Day -1).
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced greater than 60 days prior to first baseline cardiodynamic measurement (Day -1).
   * Opportunistic infections (eg, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   * Cancer or lymphoproliferative disease, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
   * Liver, kidney, heart, or other solid organ transplant.
   * Myasthenia gravis.
   * Peripheral neuropathy.
5. Has history or presence of alcoholism and/or drug abuse within the past 2 years prior to first baseline cardiodynamic measurement (Day -1), as determined by the Investigator or designee.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs.
7. Allergy to band aids, adhesive dressing, or medical tape.
8. History or presence of any of the following, deemed clinically relevant by the Investigator or designee at the screening visit or at check-in:

   * Cardiac disease; arrhythmias, presyncope, or syncopal episodes; heart failure, heart disease or risk factors for torsades de pointes (including long QT syndrome or family history of long QT syndrome).
   * Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, history of cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities.
   * Ischemic heart disease, poorly controlled hypertension, or other cardiovascular disorder
   * T wave flattening or other abnormalities which in the opinion of the Investigator or designee may interfere with the analysis of QT intervals.
   * A family history of sudden cardiac death.
9. Female participant with a positive pregnancy test at the screening visit or at check-in or who is breastfeeding and/or lactating.
10. Positive urine drug or alcohol results at the screening visit or at check-in.
11. Positive Coronavirus disease 2019 (COVID-19) result at check-in.
12. Unable to refrain from or anticipates the use of:

    * Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements, including any cytochrome P450 (CYP)3A4 inhibitors, beginning 14 days prior to the first baseline cardiodynamic measurement (Day -1).
    * Any drugs known to be inducers of CYP3A4 enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first baseline cardiodynamic measurement (Day -1). Appropriate sources (eg, Flockhart Table™) including the product label for moxifloxacin will be consulted to confirm lack of pharmacokinetic (PK)/pharmacodynamic interaction with the study drugs.
    * Any drugs known to prolong the QT/QTc interval for 28 days or 5 half-lives (whichever is longer) prior to the first baseline cardiodynamic measurement (Day -1).
13. Has been on a diet incompatible with the on study diet, in the opinion of the Investigator or designee, within the 30 days prior to first baseline cardiodynamic measurement (Day -1) and throughout the study.
14. Has made a donation of blood or had significant blood loss within 56 days prior to first baseline cardiodynamic measurement (Day -1).
15. Has made a plasma donation within 7 days prior first baseline cardiodynamic measurement (Day -1).
16. Participated in another clinical study within 30 days prior to first baseline cardiodynamic measurement (Day -1). The 30-day window will be derived from the date of the last dosing in the previous study to Day -1 of the current study.
17. Herpes infections:

    * Has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at the screening visit or check-in.
    * Has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
18. Positive results for non-herpetic viral diseases at the screening visit:

    * Hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV ribonucleic acid (RNA; nucleic acid test or polymerase chain reaction [PCR]).
    * Hepatitic B surface antigen (HBsAg+), hepatitis B virus deoxyribonucleic acid (DNA), or hepatitis B core antibody (HBcAb+) with positive hepatitis B virus DNA.
    * Human immunodeficiency virus (HIV).
19. Positive results for tuberculosis (TB) at the screening visit or has any of the following:

    * Has history of active TB infection, regardless of treatment status.
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the Investigator or designee.
    * Has evidence of latent tuberculosis infection (LTBI) as evidenced by a positive Quantiferon TB Gold (QFT) result or 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis. Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines).
    * Has had any imaging study prior to the screening visit, including x ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected Change From Baseline in QTc Interval (ΔΔQTc) for TAK-279 | Baseline, Days 1, 7, and 8
  Placebo-corrected QTc interval will be measured by continuous ECG recordings.

SECONDARY OUTCOMES:
Change From Baseline in Heart Rate (HR [ΔHR]) for TAK-279 | Baseline, Days 1, 7, and 8
  HR will be measured by continuous ECG recordings.
Change From Baseline in QTc (ΔQTc) Interval for TAK-279 | Baseline, Days 1, 7, and 8
  QTc interval will be measured by continuous ECG recordings.
Change From Baseline in PR Interval (ΔPR) for TAK-279 | Baseline, Days 1, 7, and 8
  PR interval will be measured by continuous ECG recordings.
Change From Baseline in QRS Interval (ΔQRS) for TAK-279 | Baseline, Days 1, 7, and 8
  QRS interval will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in HR (ΔΔHR) for TAK-279 | Baseline, Days 1, 7, and 8
  Placebo-corrected HR will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in ΔPR (ΔΔPR) for TAK-279 | Baseline, Days 1, 7, and 8
  Placebo-corrected PR will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in QRS (ΔΔQRS) for TAK-279 | Baseline, Days 1, 7, and 8
  Placebo-corrected QRS interval will be measured by continuous ECG recordings.
Number of Participants With Categorical Outliers for HR, PR, QRS, and QTc for TAK-279 | Baseline, Days 1, 7, and 8
  HR, PR, QRS, and QTc will be measured by continuous ECG recordings.
Change From Baseline in Electrocardiogram (ECG) Morphology for TAK-279 | Baseline, Days 1, 7, and 8
  ECG morphological analyses will be performed using the ECG waveform interpretation as defined by the central ECG laboratory's cardiologist.
Placebo-corrected Change From Baseline in QTc Interval (ΔΔQTc) for Moxifloxacin | Baseline, Days 1, 7, and 8
  Placebo-corrected QTc interval will be measured by continuous ECG recordings.
Maximum Observed Plasma Concentration (Cmax) of TAK-279 and Moxifloxacin | Days 1 (TAK-279 and Moxifloxacin) and 7 (TAK-279): Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose; Day 8 (Moxifloxacin): 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Time to Reach Cmax (tmax) of TAK-279 and Moxifloxacin | Days 1 (TAK-279 and Moxifloxacin) and 7 (TAK-279): Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose; Day 8 (Moxifloxacin): 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Area Under the Plasma Concentration-Time Curve During a Dosing Interval (tau) at Steady State (AUCτ) of TAK-279 | Days 1 and 7: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 hours (AUC0-24) of Moxifloxacin | Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose; Day 8: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESIs) | Baseline up to Day 22
Number of Participants With Markedly Abnormal Values (MAVs) in Vital signs Parameters | Baseline up to Day 9
  Vital signs assessment will include blood pressure, pulse rate, respiratory rate, and oral temperature parameters.
Number of Participants With MAVs in 12-lead ECGs Measurement | Baseline up to Day 9
  ECGs will be performed with participants in a supine position.
Number of Participants With MAVs in Clinical Laboratory Assessments | Baseline up to Day 9
  Clinical laboratory assessment will include includes hematology, chemistry, and urinalysis parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/131873ebfd4d4e1e?idFilter=%5B%22TAK-279-1001%22%5D